CLINICAL TRIAL: NCT00002625
Title: PHASE I STUDY OF TOPOTECAN AND THORACIC RADIATION
Brief Title: Topotecan and Radiation Therapy in Treating Patients With Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000063990; WCCC-CO-9492; NCI-T94-0099C; CDR0000063990 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Esophageal Cancer; Lung Cancer; Lymphoma
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent non-small cell lung cancer; recurrent adult Hodgkin lymphoma; recurrent esophageal cancer; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent small cell lung cancer; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Lymphoma; Hodgkin Disease; Carcinoma, Non-Small-Cell Lung; Lymphoma, T-Cell, Cutaneous; Small Cell Lung Carcinoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Topotecan

ARMS (1):
- Arm I (Experimental): Radiosensitization plus Radiotherapy. Topotecan hydrochloride, TOPO, NSC-609699; plus external-beam irradiation using linear accelerators with photon energies between 4 and 10 MV (electrons acceptable for the boost field).
  Interventions: Drug: topotecan hydrochloride; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Drug: topotecan hydrochloride
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
Phase I trial to study the effectiveness of topotecan and radiation therapy in treating patients who have solid tumors or lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy with radiation therapy may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Define the maximum tolerated dose and safety profile of topotecan (TOPO) administered with daily high-dose thoracic radiotherapy to a total of 60 Gy in patients with solid tumor or lymphoma.

II. Assess the qualitative and quantitative nature of the toxic effects encountered in this treatment.

III. Estimate the tissue and tumor TOPO concentrations during radiotherapy by evaluating plasma TOPO levels.

IV. Evaluate, using Western blot and immunohistochemical stain, the effects of TOPO/radiotherapy on topoisomerase I levels in peripheral blood lymphocytes (PBL).

V. Determine whether TOPO induces apoptosis in PBL from this patient population.

VI. Examine tumor tissue pre- and post-treatment (if available) for topoisomerase I levels, DNA damage, topoisomerase I/DNA complexes, and apoptotic events.

OUTLINE:

Radiosensitization plus Radiotherapy. Topotecan, TOPO, NSC-609699; plus external-beam irradiation using linear accelerators with photon energies between 4 and 10 MV (electrons acceptable for the boost field).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Microscopically confirmed solid tumor or lymphoma not potentially curable by conventional surgery or radiotherapy
* Previously unirradiated disease scheduled to receive thoracic irradiation of up to 60 Gy, including pulmonary and esophageal tumors
* No metastatic disease more effectively treated by systemic chemotherapy
* No history of brain metastases

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0 or 1
* WBC at least 4,000
* ANC at least 1,500
* Platelets at least 100,000
* Bilirubin no greater than 1.5 mg/dL
* Creatinine no greater than 1.5 mg/dL
* Calcium no greater than 11.0 mg/dL
* No pregnant or nursing women
* Pregnancy test required, as appropriate
* Effective contraception required of fertile patient

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since chemotherapy (6 weeks since nitrosoureas and mitomycin) and recovered
* At least 4 weeks since radiotherapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1995-03; Primary Completion 2000-04 (Actual); Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Forouzannia A, Schiller J, Berlin J, Hutson P, Boothman D, Storer B, Wilding G, Mehta M. A phase I study of Topotecan, as a radiosensitizer, for thoracic malignancies. Lung Cancer. 2004 Apr;44(1):111-9. doi: 10.1016/j.lungcan.2003.10.005. PMID 15013589